CLINICAL TRIAL: NCT02773407
Title: Parallel Group, Double Blinded, 1:1, Randomized Controlled Phase III Trial of Co-trimoxazole Versus Azithromycin for the Treatment of Undifferentiated Fever In Nepal
Brief Title: Nepal Undifferentiated Febrile Illness Trial
Acronym: NUFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: University of Oxford (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18NP
Record Dates: First submitted 2016-05-05; First posted 2016-05-16 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Undifferentiated Febrile Illness
Keywords: Undifferentiated febrile illness; Azithromycin; Cotrimoxazole; Efficacy; Enteric fever; Fever clearance time
MeSH Terms: conditions — Typhoid Fever | interventions — Azithromycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Azithromycin tablets 20mg/kg/day for 7 days (Maximum dose 1000mg/day)
  Interventions: Drug: Azithromycin
- Group B (Active Comparator): Co-trimoxazole tablets (Trimethoprim 10 mg/kg+Sulphamethoxazole 50 mg/kg) in two divided doses everyday for 7 days (maximum 3000mg/day)
  Interventions: Drug: Co-trimoxazole

INTERVENTIONS:
Drug: Azithromycin
  Arms: Group A
Drug: Co-trimoxazole
  Arms: Group B

SUMMARY:
The purpose of the study is to determine whether azithromycin or cotrimoxazole is the best empirical treatment for undifferentiated febrile illness in Nepal

DETAILED DESCRIPTION:
Fever is one of the most common presenting symptoms of patients presenting to health centers in Nepal. Many of the times, it is difficult to diagnose the cause of the fever by initial history, clinical examination and basic laboratory tests and the patents are treated as presumed enteric fever or fever without focus needing antimicrobials. In fact there are various causes of similarly presenting febrile illnesses including typhoid, paratyphoid, murine typhus, scrub typhus etc.

Many of the traditionally used drugs including fluoroquinolones are now resistant against enteric fever in south asia. Oral azithromycin is now commonly used to treat undifferentiated febrile illness and remains effective against enteric fever. Many physicians now also use co-trimoxazole as it was very commonly used in the treatment of enteric fever in the past. Resistance to co-trimoxazole emerged two decades ago, but has subsequently largely disappeared and nearly all Salmonella Typhi and Paratyphi A strains from Nepal are now susceptible. Anecdotal reports claim that it seems to work very well against undifferentiated febrile illness in Nepal; it is largely stocked in government health facilities and is a popular and cheap treatment option.

Both azithromycin and co-trimoxazole are available in Nepal and are extensively used in the treatment of undifferentiated febrile illness. Therefore it is important to know the better oral option to treat enteric fever and other febrile illnesses and also to have an alternative oral treatment in case resistance to azithromycin emerges.

The investigators purpose to conduct a head to head, parallel group, 1:1, double blinded randomized controlled trial to compare azithromycin and co-trimoxazole for the treatment of undifferentiated febrile illness and determine the best empirical treatment for undifferentiated febrile illness in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Fever of ≥ 38.0°C and for ≥4 days without a focus of infection
* ≥ 2 years and <65 years of age
* Able to take tablets orally
* Patient residing in Kathmandu Valley
* Able to come for follow up
* Can be reached by telephone/mobile phone 24 hours a day.
* Written informed consent to participate in the study including assent for minors in addition to parental consent.

Exclusion Criteria:

* Fever >14 days
* Pregnancy
* Obtundation
* Shock
* Visible jaundice
* Presence of signs of gastrointestinal bleeding
* History of hypersensitivity to either of the trial drugs
* Patient requiring intravenous antibiotic or hospital admission for any reason.
* Contraindication of drug for any reason (e.g. drug interactions).
* Any patient fulfilling inclusion criteria but already on antimicrobials and responding clinically to the treatment

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-08-04 (Actual); Study Completion 2019-08-04 (Actual)

PRIMARY OUTCOMES:
Fever clearance time | at least 2 days
  time from the first dose of a study drug until a temperature ≤37.5°C for at least 2 days

SECONDARY OUTCOMES:
Fever failure | over 7 days post treatment initiation
  defined by fever clearance time (FCT) >7 days post treatment initiation;
Need rescue treatment | within 63 days
  Requirement for rescue treatment as judged by the Research Medical Officer (RMO) and Attending Physician (AP)
Microbiological failure | on day 7 of treatment
  Blood culture positivity for S. Typhi or an S. Paratyphi
Relapse | within 28 days of initiation of treatment
  Culture-confirmed or syndromic enteric fever relapse
The development of any complication | within 28 days of initiation of treatment
  any complication: e.g. clinically significant bleeding, fall in the Glasgow Coma Score, perforation of the gastrointestinal tract and hospital admission
Time-to-treatment failure | within 63 days
  the time from the first dose of treatment until the date of the earliest failure event
Adverse events | within 63 days
  grade 3/4 adverse events, serious adverse events, adverse events of any grade leading to modification of study drug dose or interruption/early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Buddha Basnyat, MBBS,MSc,MD, Principal Investigator — University of Oxford
Locations (2):
- Nepal (2):
  - Nepal Civil Service Hospital, Kathmandu
  - Patan Hospital, Kathmandu

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be made available to researcher and public as a supporting material via open access journal and/or upon request by qualified research groups

REFERENCES:
- [Background] Crump JA, Kirk MD. Estimating the Burden of Febrile Illnesses. PLoS Negl Trop Dis. 2015 Dec 3;9(12):e0004040. doi: 10.1371/journal.pntd.0004040. eCollection 2015 Dec. No abstract available. PMID 26633014
- [Background] Zimmerman MD, Murdoch DR, Rozmajzl PJ, Basnyat B, Woods CW, Richards AL, Belbase RH, Hammer DA, Anderson TP, Reller LB. Murine typhus and febrile illness, Nepal. Emerg Infect Dis. 2008 Oct;14(10):1656-9. doi: 10.3201/eid1410.080236. PMID 18826840
- [Background] Thompson CN, Blacksell SD, Paris DH, Arjyal A, Karkey A, Dongol S, Giri A, Dolecek C, Day N, Baker S, Thwaites G, Farrar J, Basnyat B. Undifferentiated febrile illness in Kathmandu, Nepal. Am J Trop Med Hyg. 2015 Apr;92(4):875-878. doi: 10.4269/ajtmh.14-0709. Epub 2015 Feb 9. PMID 25667056
- [Background] Koirala S, Basnyat B, Arjyal A, Shilpakar O, Shrestha K, Shrestha R, Shrestha UM, Agrawal K, Koirala KD, Thapa SD, Karkey A, Dongol S, Giri A, Shakya M, Pathak KR, Campbell J, Baker S, Farrar J, Wolbers M, Dolecek C. Gatifloxacin versus ofloxacin for the treatment of uncomplicated enteric fever in Nepal: an open-label, randomized, controlled trial. PLoS Negl Trop Dis. 2013 Oct 31;7(10):e2523. doi: 10.1371/journal.pntd.0002523. eCollection 2013. PMID 24282626
- [Background] Arjyal A , Basnyat B, Nhan HT, Koirala S, Giri A, Joshi N, et al. A randomised controlled trial of gatifloxacin versus ceftriaxone for the treatment of uncomplicated enteric fever in Nepal. Submitted. 2015;3099(15):1-11
- [Background] Dolecek C, Tran TP, Nguyen NR, Le TP, Ha V, Phung QT, Doan CD, Nguyen TB, Duong TL, Luong BH, Nguyen TB, Nguyen TA, Pham ND, Mai NL, Phan VB, Vo AH, Nguyen VM, Tran TT, Tran TC, Schultsz C, Dunstan SJ, Stepniewska K, Campbell JI, To SD, Basnyat B, Nguyen VV, Nguyen VS, Nguyen TC, Tran TH, Farrar J. A multi-center randomised controlled trial of gatifloxacin versus azithromycin for the treatment of uncomplicated typhoid fever in children and adults in Vietnam. PLoS One. 2008 May 21;3(5):e2188. doi: 10.1371/journal.pone.0002188. PMID 18493312
- [Background] Parry CM, Ho VA, Phuong le T, Bay PV, Lanh MN, Tung le T, Tham NT, Wain J, Hien TT, Farrar JJ. Randomized controlled comparison of ofloxacin, azithromycin, and an ofloxacin-azithromycin combination for treatment of multidrug-resistant and nalidixic acid-resistant typhoid fever. Antimicrob Agents Chemother. 2007 Mar;51(3):819-25. doi: 10.1128/AAC.00447-06. Epub 2006 Dec 4. PMID 17145784
- [Background] Chinh NT, Parry CM, Ly NT, Ha HD, Thong MX, Diep TS, Wain J, White NJ, Farrar JJ. A randomized controlled comparison of azithromycin and ofloxacin for treatment of multidrug-resistant or nalidixic acid-resistant enteric fever. Antimicrob Agents Chemother. 2000 Jul;44(7):1855-9. doi: 10.1128/AAC.44.7.1855-1859.2000. PMID 10858343
- [Background] Chand HJ, Rijal KR, Neupane B, Sharma VK, Jha B. Re-emergence of susceptibility to conventional first line drugs in Salmonella isolates from enteric fever patients in Nepal. J Infect Dev Ctries. 2014 Nov 13;8(11):1483-7. doi: 10.3855/jidc.4228. PMID 25390062
- [Background] Pandit A, Arjyal A, Day JN, Paudyal B, Dangol S, Zimmerman MD, Yadav B, Stepniewska K, Campbell JI, Dolecek C, Farrar JJ, Basnyat B. An open randomized comparison of gatifloxacin versus cefixime for the treatment of uncomplicated enteric fever. PLoS One. 2007 Jun 27;2(6):e542. doi: 10.1371/journal.pone.0000542. PMID 17593957
- [Background] Arjyal A, Basnyat B, Koirala S, Karkey A, Dongol S, Agrawaal KK, Shakya N, Shrestha K, Sharma M, Lama S, Shrestha K, Khatri NS, Shrestha U, Campbell JI, Baker S, Farrar J, Wolbers M, Dolecek C. Gatifloxacin versus chloramphenicol for uncomplicated enteric fever: an open-label, randomised, controlled trial. Lancet Infect Dis. 2011 Jun;11(6):445-54. doi: 10.1016/S1473-3099(11)70089-5. Epub 2011 Apr 29. PMID 21531174
- [Derived] Giri A, Karkey A, Dangol S, Arjyal A, Pokharel S, Rijal S, Gajurel D, Sharma R, Lamsal K, Shrestha P, Prajapati G, Pathak S, Shrestha SR, K C RK, Pandey S, Thapa A, Shrestha N, Thapa RK, Poudyal B, Phuong DNT, Baker S, Kestelyn E, Geskus R, Thwaites G, Basnyat B. Trimethoprim-sulfamethoxazole Versus Azithromycin for the Treatment of Undifferentiated Febrile Illness in Nepal: A Double-blind, Randomized, Placebo-controlled Trial. Clin Infect Dis. 2021 Oct 5;73(7):e1478-e1486. doi: 10.1093/cid/ciaa1489. PMID 32991678
- [Derived] Pokharel S, Basnyat B, Arjyal A, Mahat SP, Kc RK, Bhuju A, Poudyal B, Kestelyn E, Shrestha R, Phuong DNT, Thapa R, Karki M, Dongol S, Karkey A, Wolbers M, Baker S, Thwaites G. Co-trimoxazole versus azithromycin for the treatment of undifferentiated febrile illness in Nepal: study protocol for a randomized controlled trial. Trials. 2017 Oct 2;18(1):450. doi: 10.1186/s13063-017-2199-6. PMID 28969659